CLINICAL TRIAL: NCT02080767
Title: Clinical Protocol to Treat Individuals With Tecovirimat (ST-246) After Exposure to Orthopox Viruses
Brief Title: Tecovirimat (ST-246) Treatment for Orthopox Virus Exposure
Status: Available | Type: Expanded Access
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: M-10331; S-11-10 (Other: Sponsor)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Smallpox; Monkeypox
MeSH Terms: conditions — Smallpox; Mpox, Monkeypox | interventions — tecovirimat

INTERVENTIONS:
Drug: Tecovirimat — Oral tablet 600mg daily dose(three capsules, 200 mg/capsule)
  Other Names: ST 246

SUMMARY:
The purpose of this clinical protocol is to treat individuals with Tecovirimat after exposure to orthopox viruses.

DETAILED DESCRIPTION:
Rationale: Tecovirimat (TPOXX) is approved by FDA for treatment of smallpox. However, the therapeutic human dose for treatment of orthopox virus infections or a significant adverse reaction to vaccinia resulting from vaccination, secondary transmission, or other exposure, has not yet been fully established.

Treatment: Based on the interpretation of currently available animal efficacy and human safety and PK data, the proposed human adult or pediatric patient (≥ 40 kg) therapeutic regimen is 600 mg (3 capsules of 200 mg) orally twice daily (BID) for at least 14 days, taken 30 minutes after a meal consisting of about 600 calories and 30% (25 grams) fat, which is the same as treatment for smallpox. If a dose is missed it should be taken as soon as possible unless it is near the next dose time. Doses should not be doubled in the event of a missed dose. Treatment may be extended beyond 14 days, with sponsor approval, if the investigator deems necessary. Nonclinical safety data support use for up to 90 days.

The pediatric dosing recommendation is derived from the TPOXX package insert based on the body weight: 200 mg twice daily for patients of 13-25kg (29-45pounds); 400 mg twice daily for patients 25-40kg (55-87pounds) and 600 mg twice daily for pediatric patients over 40kg (88pounds)

Clinical Evaluation: Medical history and concomitant medications will be recorded, and a physical examination with vital signs [eg, body weight, blood pressure, heart rate, respiratory rate, temperature, and height (only once)] will be completed. Photographs of affected areas, should lesions develop, may be taken. Patients will be followed for at least 30 days after receiving the last tecovirimat dose or until their infection improves.

ELIGIBILITY:
Inclusion Criteria:

* DoD-affiliated personnel (including US civilian employees, contractors and other US personnel and dependents, as well as allied military forces and local nationals) of any age, not breastfeeding
* Has been exposed to or infected with orthopox viruses (ie, variola (smallpox), vaccinia, monkeypox, or cowpox) OR Has developed serious complications from vaccinia vaccination (eg, eczema vaccinatum, progressive vaccinia, generalized vaccinia that is severe or persistent, and select cases of inadvertent inoculation due to severe pain related to mucosal involvement, ocular involvement) resulting from vaccination, secondary transmission, or other exposure
* Is available for clinical follow-up for duration of the treatment and follow-up period
* Must be able to swallow capsules

Exclusion Criteria:

* Has hypersensitivity to tecovirimat
* Unable or unwilling to cooperate with the requirements of the treatment protocol
* Breast-feeding patients. Note that breast-feeding females will be counseled that tecovirimat has not been studied in breast-feeding women and may opt to cease breast-feeding for the duration of the treatment and at least 30 days after the last dose of drug and thus be eligible for enrollment. Women who choose to continue breast-feeding will not be enrolled in this treatment protocol.

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] Hatmal MM, Al-Hatamleh MAI, Olaimat AN, Ahmad S, Hasan H, Ahmad Suhaimi NA, Albakri KA, Abedalbaset Alzyoud A, Kadir R, Mohamud R. Comprehensive literature review of monkeypox. Emerg Microbes Infect. 2022 Dec;11(1):2600-2631. doi: 10.1080/22221751.2022.2132882. PMID 36263798